CLINICAL TRIAL: NCT04448717
Title: Seroprevalence of SARS-CoV-2 Antibodies and Development of Immunity in a Public School Population - a Population-based Observational Study to Inform Policy Making
Brief Title: COVID-19: Longitudinal Study of Seroprevalence of SARS-CoV-2 Antibodies and Development of Immunity in School Children
Acronym: CiaoCorona
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss School of Public Health (SSPH+) (Other)
Responsible Party: Principal Investigator, Susi Kriemler, Prof. Dr. med., University of Zurich
Other Study IDs: 2020-01336
Record Dates: First submitted 2020-06-18; First posted 2020-06-26 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: SARS-CoV 2; COVID-19
Keywords: Seroprevalence; Seroepidemiology; School children; Switzerland; Schools; Households; Students
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serological Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum and serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Children and adolescents: Children and adolescents in primary and secondary schools (aimed sample size: 2500)
  Interventions: Diagnostic Test: COVID-19 Antibody testing
- Parents: Parents of participating children (aimed sample size: 3000)
  Interventions: Diagnostic Test: COVID-19 Antibody testing
- School personnel: School personnel (teaching, administrative, maintenance, etc.) (aimed sample size: 2500)
  Interventions: Diagnostic Test: COVID-19 Antibody testing

INTERVENTIONS:
Diagnostic Test: COVID-19 Antibody testing — COVID-19 Antibody testing in venous blood and/or saliva samples.

SUMMARY:
There is a lack of knowledge about how many children are infected with SARS-CoV-2, how often they are asymptomatic, and how long the immunity persists.

The main purpose of this study is to measure antibodies to SARS-CoV-2, symptoms, and risk factors in a representative cohort of children and adolescents in the canton of Zurich, Switzerland, shortly after re-opening of the school system and thereafter. The study also investigates antibodies to SARS-CoV-2 in parents of the children and school personnel.

DETAILED DESCRIPTION:
The role of children and adolescents in the transmission of SARS-CoV-2 remains highly unclear and has been a key question since the early days of the pandemic. It has important consequences for policy decisions, especially concerning the opening of the schools, sport facilities and intergenerational contacts. However, the information on true infection rate and seroprevalence of SARS-CoV-2 is not known in children in Switzerland (and globally), as testing was limited to risk groups and those with SARS-CoV-2 coronavirus disease 2019 (COVID-19) related symptoms. In addition, indications for testing were not uniform and handled heterogeneously. Hence, it is not known whether children are less frequently infected or simply less symptomatic.

This study builds up a system to monitor the seroprevalence of SARS-CoV-2 in children and adolescents who attend school in the canton of Zürich, Switzerland. The investigators aim to assess children of randomly selected primary and secondary schools during the first weeks of re-entering school from all districts of the canton of Zurich in June and July 2020, after the temporary closure due to COVID-19 pandemic, and again in October/November 2020, February/March 2021, November/December 2021, and again in the second half of 2022. The detailed time plan including possible further assessments will be defined depending on the evolution of the pandemic (e.g., 2023). A follow-up capturing health status, symptoms and behaviors over time is important, since it is currently under investigation whether persons may be at risk for reinfection. Thus, a longitudinal assessment is crucial to determine the extent and duration of immunity.

In addition, the seroprevalence of SARS-CoV-2 in the parents of the participating children will be tested in August/September 2020, to examine clusters of infections in households. Seroprevalence of SARS-CoV-2 in school personnel will be tested in August/September 2020 and subsequently in October/November 2020 and February/March 2021, to examine temporal changes in the seroprevalences in the whole school community. Further testing of adults is not planned.

In different subpopulations, further in-depth analysis of immunity markers will be performed in the future.

This study complements the ongoing coordinated efforts of seroprevalence studies in adults in Switzerland, through the Swiss School of Public Health (SSPH+) coordinated CORONA IMMUNITAS studies.

ELIGIBILITY:
Inclusion Criteria:

* Any school child residing in Switzerland aged 5 years or older and attending a consenting to participate public or private school that hosts classes of interest (grade 1 through 9) in the canton of Zürich.
* Parents of participating children.
* Personnel employed in the participating schools.
* No acute respiratory and SARS-CoV-2 infection:

  * In case of unknown respiratory infection, no presence of symptoms for at least 48 hours.
  * In case of confirmed SARS-CoV-2 infection: inclusion at the earliest 21 days from PCR-positive diagnosis after the onset of potential symptoms and no presence of symptoms for at least 48 hours (according to Standard of Care).
* Informed consent of parents or legal guardians and children, or the adult participant.

Exclusion Criteria:

* No informed consent by schools or children, or the adult participant.
* Schools with <40 students in one of the sampled grades (1, 2, 4, 5, 7, or 8).
* Children of Kindergarten age and younger.
* Suspicion of acute COVID-19 infection.
* Special need schools.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: School children, attending grades 1 to 9 in a public or private school in the Canton of Zurich, Switzerland.
  Parents of participating children. School personnel of participating schools.
Sampling Method: Probability Sample
Enrollment: 4250 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Seroprevalence of SARS-CoV-2 IgG, IgM and/or IgA antibodies | at inclusion
  Seroprevalence of SARS-CoV-2 IgG, IgM and/or IgA antibodies in randomly selected 5- to 16-year-old population of school-children, their parents, and school personnel, after the peak phase of the first major wave shortly after re-opening of schools in the canton of Zürich, Switzerland.
Seroprevalence of SARS-CoV-2 IgG, IgM and/or IgA antibodies | Month 4-5
  Seroprevalence of SARS-CoV-2 IgG, IgM and/or IgA antibodies in randomly selected 5- to 16-year-old population of school-children and school personnel after 4-5 after recruitement in the canton of Zürich, Switzerland.
Seroprevalence of SARS-CoV-2 IgG, IgM and/or IgA antibodies | Month 8-9
  Seroprevalence of SARS-CoV-2 IgG, IgM and/or IgA antibodies in randomly selected 5- to 16-year-old population of school-children and school personnel after 8-9 months after recruitment in the canton of Zürich, Switzerland.
Seroprevalence of SARS-CoV-2 IgG antibodies | Month 17-18
  Seroprevalence of SARS-CoV-2 IgG antibodies in randomly selected 5- to 16-year-old population of school-children and school personnel after 17-18 months after recruitment in the canton of Zürich, Switzerland.
Seroprevalence of SARS-CoV-2 IgG antibodies | Month 24-30
  Seroprevalence of SARS-CoV-2 IgG antibodies in randomly selected 5- to 16-year-old population of school-children and school personnel after 24-30 months after recruitment in the canton of Zürich, Switzerland.

SECONDARY OUTCOMES:
Presence of self-reported symptoms | at inclusion
  Presence of symptoms (from January 2020) suggestive of a common cold, influenza and similar upper respiratory tract infections prior to the first study visit.
Proportion of seropositive children reporting COVID-19 related symptoms from January 2020 | at inclusion
  Proportion of seropositive children reporting symptoms suggestive of a common cold, influenza and similar upper respiratory tract infections between January 2020 and first study visit.
Presence of self-reported symptoms | within 36 months of follow-up
  Presence of symptoms (from January 2020) suggestive of a common cold, influenza and similar upper respiratory tract infections during the follow-up.
Incidence of symptoms in initially seropositive participants | within 36 months of follow-up
  Incidence of self-reported symptoms and SARS-CoV-2 infections after the first study visit in initially seropositive participants.
Proportion of participants, seronegative at inclusion, with symptoms in the follow-up | within 36 months of follow-up
  Proportion of seronegative participants of the first investigation wave who will self-report symptoms and infection with SARS-CoV-2.
Presence of risk factors for infection at inclusion (assessment via custom questionnaire) | at inclusion
  Potential personal (socioeconomic characteristics, health status, presence of infection in family, personal hygiene and social distancing measures) and school-level (implementation of informational, social distancing and hygiene measures at school) risk and preventive factors for SARS-CoV-2 infection prior to the study. Questionnaire includes HBSC and custom questions.
Presence of risk factors for infection during follow-up (assessment via custom questionnaire) | within 36 months of follow-up
  Potential personal (socioeconomic characteristics, health status, presence of infection in family, personal hygiene and social distancing measures) and school-level (implementation of informational, social distancing and hygiene measures at school) risk and preventive factors for SARS-CoV-2 infection during the follow-up. Questionnaire includes HBSC and custom questions.
Self-reported lifestyle changes of participants at inclusion | at inclusion
  Changes in lifestyle during the lock-down, compared to prior to it: frequency and duration (in hours, daily) of physical activity, duration (in hours, daily) of sleep, duration of screen-based media-use (in hours, daily). This outcome is measured only in the children population.
Self-reported lifestyle changes of participants during follow-up | within 36 months of follow-up
  Changes in lifestyle after the lock-down and school reopening, compared to during lock-down: frequency and duration (in hours, daily) of physical activity, duration (in hours, daily) of sleep, duration of screen-based media-use (in hours, daily). This outcome is measured only in the children population.
Self-reported mental well-being (KINDL questionnaire) | within 36 months of follow-up
  Changes over the study time in mental well-being of the participants during and after the lock-down: frequency scale (never/rarely/sometimes/often/always) of self-reported stress, anxiety, self-confidence feelings in the last 7 days. This outcome is measured only in the children population.
Self-reported mental well-being (HBSC questionnaire) | within 36 months of follow-up
  Changes over the study time in mental well-being of the participants during and after the lock-down: frequency scale (daily/weekly/monthly/rarer) of self-reported sadness, anxiety and sleeping problems (HBSC questionnaire question on mental well-being). This outcome is measured only in the children population.
Self-reported quality of life (KINDL questionnaire) | within 36 months of follow-up
  Changes over the study time in quality-of-life of the participants during and after the lock-down: frequency scale (never/rarely/sometimes/often/always) assessment of self-reported positive and negative social interactions with family, friends and in the school environment in the last 7 days. This outcome is measured only in the children population.
Prevalence of seropositive SARS-Cov-2 clusters in schools at inclusion | at inclusion
  Prevalence of clusters of seropositive children, adolescents, and school personnel within schools and classes at baseline.
Incidence of seropositive SARS-Cov-2 clusters in schools during the follow-up | within 36 months of follow-up
  Incidence of clusters of seropositive children, adolescents, and school personnel within schools and classes during the follow-up.
Change in seropositive participants within school or class, depending on the initial proportion of seropositive participants | within 36 months of follow-up
  Impact of the number of children/adolescents and school personnel at a specific period (baseline, at the second and third testing date) within a school or class to the subsequent seropositivity within the same group.
Effect of risk factors and preventive measures on SARS-CoV-2 infection incidence within schools | within 36 months of follow-up
  Incidence of seropositive children and school personnel according to potential risk factors and preventive measures for SARS-CoV-2 infection within schools.

OTHER OUTCOMES:
Evolution of cellular immunity over time | within 36 months of follow-up
  Cellular immunity (T & B cells) in a subsample of previously antibody positive and antibody negative (controls) children.
Long COVID | within 36 months of follow-up
  Self-reported symptoms compatible with Long COVID (i.e., >3months) in seropositive versus seronegative children. Symptoms adapted from International Severe Acute Respiratory and emerging Infection Consortium (ISARIC).

CONTACTS AND LOCATIONS:
Overall Officials: Susi Kriemler, Prof., Principal Investigator — University of Zurich
Locations (1):
- Epidemiology, Biostatistics and Prevention Institute (EBPI), University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Sensitive clinical data from vulnerable population (children) will be collected. Therefore, it is not yet decided, if it will be possible to share IPD while preserving participant autonomy and privacy.

REFERENCES:
- [Background] Ulyte A, Radtke T, Abela IA, Haile SR, Berger C, Huber M, Schanz M, Schwarzmueller M, Trkola A, Fehr J, Puhan MA, Kriemler S. Clustering and longitudinal change in SARS-CoV-2 seroprevalence in school children in the canton of Zurich, Switzerland: prospective cohort study of 55 schools. BMJ. 2021 Mar 17;372:n616. doi: 10.1136/bmj.n616. PMID 33731327
- [Background] Radtke T, Ulyte A, Puhan MA, Kriemler S. Long-term Symptoms After SARS-CoV-2 Infection in Children and Adolescents. JAMA. 2021 Jul 15;326(9):869-71. doi: 10.1001/jama.2021.11880. Online ahead of print. PMID 34264266
- [Background] Ammann P, Ulyte A, Haile SR, Puhan MA, Kriemler S, Radtke T. Perceptions towards mask use in school children during the SARS-CoV-2 pandemic: descriptive results from the longitudinal Ciao Corona cohort study. Swiss Med Wkly. 2022 Apr 20;152:w30165. doi: 10.4414/smw.2022.w30165. eCollection 2022 Apr 11. PMID 35748765
- [Background] Peralta GP, Camerini AL, Haile SR, Kahlert CR, Lorthe E, Marciano L, Nussbaumer A, Radtke T, Ulyte A, Puhan MA, Kriemler S. Lifestyle Behaviours of Children and Adolescents During the First Two Waves of the COVID-19 Pandemic in Switzerland and Their Relation to Well-Being: An Observational Study. Int J Public Health. 2022 Sep 8;67:1604978. doi: 10.3389/ijph.2022.1604978. eCollection 2022. PMID 36158782
- [Background] Blankenberger J, Haile SR, Puhan MA, Berger C, Radtke T, Kriemler S, Ulyte A. Prediction of Past SARS-CoV-2 Infections: A Prospective Cohort Study Among Swiss Schoolchildren. Front Pediatr. 2021 Aug 16;9:710785. doi: 10.3389/fped.2021.710785. eCollection 2021. PMID 34485200
- [Background] Ulyte A, Radtke T, Abela IA, Haile SR, Braun J, Jung R, Berger C, Trkola A, Fehr J, Puhan MA, Kriemler S. Seroprevalence and immunity of SARS-CoV-2 infection in children and adolescents in schools in Switzerland: design for a longitudinal, school-based prospective cohort study. Int J Public Health. 2020 Dec;65(9):1549-1557. doi: 10.1007/s00038-020-01495-z. Epub 2020 Oct 15. PMID 33063141
- [Background] Haile SR, Gunz S, Peralta GP, Ulyte A, Raineri A, Rueegg S, Yasenok V, Radtke T, Puhan MA, Kriemler S. Health-Related Quality of Life and Adherence to Physical Activity and Screen Time Recommendations in Schoolchildren: Longitudinal Cohort Ciao Corona. Int J Public Health. 2023 Jul 19;68:1606033. doi: 10.3389/ijph.2023.1606033. eCollection 2023. PMID 37538234
- [Background] Haile SR, Peralta GP, Raineri A, Rueegg S, Ulyte A, Puhan MA, Radtke T, Kriemler S. Determinants of health-related quality of life in healthy children and adolescents during the COVID-19 pandemic: Results from a prospective longitudinal cohort study. Eur J Pediatr. 2024 May;183(5):2273-2283. doi: 10.1007/s00431-024-05459-w. Epub 2024 Feb 27. PMID 38411717
- [Background] Haile SR, Raineri A, Rueegg S, Radtke T, Ulyte A, Puhan MA, Kriemler S. Heterogeneous evolution of SARS-CoV-2 seroprevalence in school-age children: Results from the school-based cohort study Ciao Corona in November-December 2021 in the canton of Zurich. Swiss Med Wkly. 2023 Jan 30;153:40035. doi: 10.57187/smw.2023.40035. PMID 36787493
- [Background] Ulyte A, Radtke T, Abela IA, Haile SR, Blankenberger J, Jung R, Capelli C, Berger C, Frei A, Huber M, Schanz M, Schwarzmueller M, Trkola A, Fehr J, Puhan MA, Kriemler S. Variation in SARS-CoV-2 seroprevalence across districts, schools and classes: baseline measurements from a cohort of primary and secondary school children in Switzerland. BMJ Open. 2021 Jul 26;11(7):e047483. doi: 10.1136/bmjopen-2020-047483. PMID 34312201
- [Background] Kriemler S, Ulyte A, Ammann P, Peralta GP, Berger C, Puhan MA, Radtke T. Surveillance of Acute SARS-CoV-2 Infections in School Children and Point-Prevalence During a Time of High Community Transmission in Switzerland. Front Pediatr. 2021 Mar 16;9:645577. doi: 10.3389/fped.2021.645577. eCollection 2021. PMID 33796490
- [Result] Raineri A, Radtke T, Rueegg S, Haile SR, Menges D, Ballouz T, Ulyte A, Fehr J, Cornejo DL, Pantaleo G, Pellaton C, Fenwick C, Puhan MA, Kriemler S. Persistent humoral immune response in youth throughout the COVID-19 pandemic: prospective school-based cohort study. Nat Commun. 2023 Nov 27;14(1):7764. doi: 10.1038/s41467-023-43330-y. PMID 38012137
- [Derived] Raineri A, Rueegg S, Zimmermann P, Regamey N, Benden C, Haile SR, Ulyte A, Puhan MA, Kriemler S, Radtke T. Long COVID in children and adolescents: results from three cross-sectional school-based cohorts with adjudication. Swiss Med Wkly. 2025 Oct 20;155:4337. doi: 10.57187/s.4337. PMID 41114667
- [Derived] Haile SR, Peralta GP, Adams M, Bharadwaj AN, Bassler D, Moeller A, Natalucci G, Radtke T, Kriemler S. Health-related quality of life in children and adolescents born very preterm and its correlates: a cross-sectional study. BMJ Paediatr Open. 2024 Oct 10;8(1):e002885. doi: 10.1136/bmjpo-2024-002885. PMID 39389623